CLINICAL TRIAL: NCT06052904
Title: mHealth-delivered Music Breathing Therapy to Enhance Resilience and Improve Quality of Life of Caregivers of Children Newly Diagnosed With Cancer: A Pilot Randomized Controlled Trial
Brief Title: Music Breathing for Caregivers of Children Newly Diagnosed With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Tan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAED-2022-024
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Oncology; Psychological Distress
Keywords: Music breathing; Cancer; Caregivers; Children; Psychological distress; Resilience
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Home-based music breathing therapy comprising eight 1-hour weekly sessions for 2 months delivered through Zoom, an online video conferencing platform, by a qualified music therapist.
  Interventions: Behavioral: mHealth-delivered music breathing therapy
- Control group (Active Comparator): Eight weekly online educational modules on medical information and advice about caring for a child who has been newly diagnosed with cancer via email for 2 months.
  Interventions: Behavioral: Online educational modules

INTERVENTIONS:
Behavioral: mHealth-delivered music breathing therapy — Parental caregivers in the intervention group will receive individual home-based music breathing therapy comprising eight 1-hour weekly sessions for 2 months delivered through Zoom, by a qualified music therapist based on a standardized and validated music breathing instruction manual. The music breathing therapy comprises four breathing phases, namely "Discovery Breathing", "Triangular Breathing", "Silent Breathing", and "Music Breathing". In each session, participants will practice breathing for approximately 20-25 minutes in silence or with music in a sitting position. Thereafter, the participants will be instructed to create a Mandala drawing to visualize the effects of breathing on their mental body image, emotions, and thoughts. Each session will end with a debriefing session, which will serve to verbally integrate and reflect the participants' experiences and mental states.
  Arms: Intervention group
Behavioral: Online educational modules — Participants in the control group will receive eight weekly online educational modules via email for 2 months. The content of the online educational modules will include medical information and advice about caring for a child who has been newly diagnosed with cancer.
  Arms: Control group

SUMMARY:
This proposed pilot randomised controlled trial aims to examine the effect of mobile health-delivered music breathing therapy in enhancing resilience, reducing psychological distress and caregiver strain, and improving the coping and quality of life of parental caregivers of children newly diagnosed with cancer.

DETAILED DESCRIPTION:
Parents of children with cancer experience considerable stress and distress from the time of their child's life-threatening diagnosis. Music therapy, for example, music breathing therapy, has been increasingly used as a nonpharmacological care strategy in the healthcare field. Music breathing therapy is an adaptation of the Bonny Method of Guided Imagery and Music. It has demonstrated promising potential for enhancing resilience and alleviating psychological distress among diverse populations, including women with complex post-traumatic stress disorder, individuals with work-related stress and caregivers of dementia patients. However, it is unclear whether this is a feasible and acceptable approach to enhance resilience, reduce psychological distress, and improve the quality of life of Chinese caregivers of children newly diagnosed with cancer.

Aims:

* To assess the effects of a mobile health-delivered music breathing therapy in enhancing resilience, reducing psychological distress (i.e., depression, anxiety, and stress) and caregiver strain, and improving coping and quality of life of parental caregivers of children newly diagnosed with cancer
* To determine the feasibility (in terms of recruitment rates, dropout rates, engagement rates, randomization process, and intervention delivery mode), and acceptability of the intervention.

Hypotheses:

It is hypothesized that compared with caregivers who receive usual care, those who receive the mHealth-delivered music breathing therapy will report higher levels of resilience (primary outcome), lower levels of psychological distress (i.e., depression, anxiety, and stress) and caregiver strain, better coping and quality of life at the 2-month (immediately after intervention) and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

Parental caregivers (the primary caregiver; either mother or father) who

* has a child (aged under 19 years) who has been diagnosed with cancer at least 2 months but not more than 12 months prior.
* can read and communicate in Chinese (Cantonese or Mandarin)
* has Internet access through any mobile device (e.g., a cell phone, tablet or laptop with camera and microphone features).
* is willing to download and use Zoom as the intervention delivery platform.

Exclusion Criteria:

* has a child who has been diagnosed with cancer and has major comorbid conditions and/or who is receiving end-of-life care.
* is caring for more than one child with a chronic or critical illness or caring for another family member with a chronic illness.
* is currently participating in any interventions or additional counselling services.
* has a diagnosed mental illness, cognitive impairment or learning problem, and/or is taking regular psychotropic medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Resilience | 2-month after baseline (immediately after the intervention)
  The Chinese version of the Connor-Davidson Resilience Scale will be used to assess the caregivers' levels of resilience. This scale consists of 25 items, rated on a 5-point Likert scale from 0 (not true at all) to 4 (true nearly all of the time). A higher total score indicates higher level of resilience.
Resilience | 6-month after baseline
  The Chinese version of the Connor-Davidson Resilience Scale will be used to assess the caregivers' levels of resilience. This scale consists of 25 items, rated on a 5-point Likert scale from 0 (not true at all) to 4 (true nearly all of the time). A higher total score indicates a higher level of resilience.

SECONDARY OUTCOMES:
Psychological distress (i.e., depression, anxiety and stress) | 2-month and 6-month after baseline
  The Chinese version of the 21-item Depression Anxiety Stress Scale will be used to measure caregivers' mental health states of depression, anxiety, and stress over the past week. It is a set of three self-report scales, each of which comprises 7 items, rated on a 4-point Likert scale from 0 (did not apply at all over the last week) to 3 (applied very much or most of the time); a higher total score indicates a greater level of depression, anxiety and/or stress.
Caregiver strain | 2-month and 6-month after baseline
  The Chinese version of the Modified Caregivers Strain Index will be used to assess the caregiver strain of the participants. Items rated on a 3-point Likert scale (0=no, 1=yes, sometimes, and 2=yes, always); a higher total score indicates a higher level of strain experienced by the caregiver.
Coping response | 2-month and 6-month after baseline
  The Chinese version of the Brief Coping Orientation to Problems Experienced Inventory will be used to evaluate the coping responses of the parental caregivers. Items rated on a 4-point Likert scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot); a higher total score indicates a greater utilization of that specific type of coping strategy.
Caregiver's quality of life | 2-month and 6-month after baseline
  World Health Organization Quality-of-Life Scale will be used to evaluate the quality of life of caregivers. Items are rated on a 5-point Likert scale from 1 to 5; a higher total score indicates a higher quality of life.
Feasibility outcomes - recruitment rate | Change from recruitment to 6-month follow-up
  Recruitment rates will be calculated as the number of participants who consented to participate in the study divided by the number of participants who meet the inclusion criteria.
Feasibility outcomes - intervention engagement/adherence rate | Change from recruitment to 6-month follow-up
  Intervention engagement/adherence will be calculated as the number of participants who have completed the music breathing sessions and follow-up sessions, as well as spending at least once daily in performing self-practice music breathing throughout the 2-month intervention period, divided by the number of intervention group participants who have completed the study.
Feasibility outcomes - Retention rate | Change from recruitment to 6-month follow-up
  Retention rate will be calculated as the number of participants who have completed the study divided by the number of randomised participants.
Acceptability - Satisfaction | 2-month follow-up (immediately after intervention)
  Caregivers' perceived satisfaction will be assessed using an 12-item investigator-designed satisfaction survey, a higher total score indicates a higher level of satisfaction.
Acceptability | 2-month follow-up (immediately after intervention)
  A semi-structured individual interview will be used to explore participants' perceptions and experiences of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ankie Tan Cheung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No